CLINICAL TRIAL: NCT03546842
Title: A Phase III Open-label Safety and Immunogenicity Study of GARDASIL™9 Administered to 9- to 26-Year-Old Females and Males in Vietnam
Brief Title: Safety and Immunogenicity Study of V503 (GARDASIL™9, 9vHPV Vaccine) Administered to 9- to 26-Year-Old Females and Males in Vietnam (V503-017)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V503-017; 2017-001205-33 (EudraCT Number); V503-017 (Other: Merck Protocol Number)
Record Dates: First submitted 2018-05-23; First posted 2018-06-06 (Actual); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Papillomavirus Infections; Uterine Cervical Neoplasms; Vulvar Neoplasms; Vaginal Neoplasms; Adenocarcinoma in Situ; Condylomata Acuminata
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms; Vulvar Neoplasms; Vaginal Neoplasms; Adenocarcinoma in Situ; Condylomata Acuminata

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- 9vHPV vaccine (Experimental): Participants will receive a single 0.5-mL intramuscular injection of the 9vHPV vaccine at Day 1, Month 2, and Month 6
  Interventions: Biological: 9vHPV vaccine

INTERVENTIONS:
Biological: 9vHPV vaccine — 9-valent HPV [Types 6, 11, 16, 18, 31, 33, 45, 52, and 58] L1 virus-like particle vaccine in a 0.5-mL intramuscular injection
  Other Names: V503; GARDASIL™9

SUMMARY:
This study will evaluate the safety and immunogenicity of V503 (GARDASIL™9, 9vHPV vaccine) administered to 9- to 26-year-old females and males in Vietnam. The study hypothesis states that V503 induces acceptable anti-human papillomavirus (HPV) 6, 11, 16, 18, 31, 33, 45, 52, and 58 seroconversion at 4 weeks postdose 3.

ELIGIBILITY:
Inclusion Criteria:

* In good physical health
* Participants 9 to 15 years of age: has not had coitarche and do not plan on becoming sexually active during the study
* Participants 16 to 26 year of age: has never had Papanicolaou (Pap) testing or has had only normal Pap test results. Has a lifetime history of ≤4 male and/or female sexual partners.
* Female participants 16 to 26 years of age: has not had sex with males or has had sex with males and used effective contraception, and understands and agrees that during the study she should not have sexual intercourse with males without effective contraception (rhythm method, withdrawal, and emergency contraception are not acceptable methods of contraception per-protocol).

Exclusion Criteria:

* Known allergy to any vaccine component, including aluminum, yeast, or BENZONASE™
* History of severe allergic reaction that required medical intervention
* Has thrombocytopenia or any coagulation disorder that would contraindicate intramuscular injections
* Concurrently enrolled in clinical studies of investigational agents
* Immunocompromised or has been diagnosed with congenital or acquired immunodeficiency, human immunodeficiency virus (HIV) infection, lymphoma, leukemia, systemic lupus erythematosus, rheumatoid arthritis, juvenile rheumatoid arthritis, inflammatory bowel disease, or other autoimmune condition
* Had a splenectomy
* User of recreational or illicit drugs or has had a recent history (within the last year) of drug abuse or dependence. Alcohol abusers are defined as those who drink despite recurrent social, interpersonal, and/or legal problems as a result of alcohol use.
* History of a positive test for HPV
* Male participants 16 to 26 years of age: history of HPV-related external genital lesions (e.g., condyloma acuminata) or HPV-related anal lesions (e.g., condyloma acuminata, or anal intraepithelial neoplasia) or anal cancer.
* Female participants 16 to 26 years of age: history of an abnormal cervical biopsy result (showing cervical intraepithelial neoplasia or worse).
* Female participants 16 to 26 years of age: history of HPV-related external genital lesions (e.g., condyloma acuminata, or vulvar intraepithelial neoplasia) or external genital cancer, HPV-related vaginal lesions (e.g., condyloma acuminata, or vaginal intraepithelial neoplasia) or vaginal cancer, or HPV-related anal lesions (e.g., condyloma acuminata, or anal intraepithelial neoplasia) or anal cancer.
* Female participants: pregnant as determined by a serum pregnancy test or urine pregnancy test that is sensitive to 25 mIU/mL beta human chorionic gonadotropin (β-hCG).
* Female participants: expecting to donate eggs during the study.
* Receiving or has received a prohibited immunosuppressive therapy in the year prior to the study
* Received any immune globulin product or blood-derived product within the 3 months prior to the Day 1 vaccination, or plans to receive any such product during the study
* Received inactivated or recombinant vaccines within 14 days prior to the Day 1 vaccination or has received live vaccines within 21 days prior to the Day 1 vaccination
* Received a marketed HPV vaccine, or has participated in an HPV vaccine clinical study and has received either active agent or placebo
* Is or has an immediate family member (e.g., spouse, parent/legal guardian, sibling or child) who is investigational site or sponsor staff directly involved with this study.

Ages: 9 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 201 (Actual)
Dates: Start 2018-06-29 (Actual); Primary Completion 2019-01-29 (Actual); Study Completion 2019-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- National Institute of Hygiene and Epidemiology ( Site 0001), Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Thiem VD, Quang ND, Tuan NH, Cheon K, Gallagher N, Luxembourg A, Group T, Badshah C. Immunogenicity and safety of a nine-valent human papillomavirus vaccine in Vietnamese males and females (9 to 26 years of age): an open-label, phase 3 trial. Hum Vaccin Immunother. 2021 Jul 3;17(7):1980-1985. doi: 10.1080/21645515.2020.1865739. Epub 2021 Apr 12. PMID 33844623

RESULTS

PARTICIPANT FLOW:
Groups:
- 9vHPV Vaccine: Participants received a single 0.5-mL intramuscular injection of the 9-valent human papillomavirus (9vHPV) vaccine at Day 1, Month 2, and Month 6
Period: Overall Study
Arm/Group | 9vHPV Vaccine
Started | 201
Vaccination 1 | 200
Vaccination 2 | 200
Vaccination 3 | 198
Completed | 198
Not Completed | 3
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- 9vHPV Vaccine: Participants received a single 0.5-mL intramuscular injection of the 9vHPV vaccine at Day 1, Month 2, and Month 6
Arm/Group | 9vHPV Vaccine
Number analyzed (Participants) | 201
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.8 (4.4) [lower limit 4.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135
  Male | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 201
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 201
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Seroconversion Percentages to HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58 at Month 7
Description: Seroconversion was defined as a participant who was anti-HPV seronegative at Day 1 and became seropositive at 4 weeks postdose 3 (Month 7). Anti-HPV antibodies were measured using a Competitive Luminex Immunoassay.
Time Frame: 4 weeks postdose 3 (Month 7)
Population: All allocated participants who were seronegative to the appropriate HPV type at Day 1, received all 3 vaccinations with the correct dose within acceptable day ranges, provided a serum sample within 21 to 49 days postdose 3, and had no protocol deviations that could interfere with the evaluation of participant's immune response to 9vHPV vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 9vHPV Vaccine
Number analyzed (Participants) | 195
Percentage of Participants
  Anti-HPV 6: number analyzed (Participants) | 190
  Anti-HPV 6 | 100 [98.1 to 100.0]
  Anti-HPV 11: number analyzed (Participants) | 190
  Anti-HPV 11 | 100 [98.1 to 100.0]
  Anti-HPV 16: number analyzed (Participants) | 187
  Anti-HPV 16 | 100 [98.0 to 100.0]
  Anti-HPV 18: number analyzed (Participants) | 190
  Anti-HPV 18 | 100.0 [98.1 to 100.0]
  Anti-HPV 31: number analyzed (Participants) | 188
  Anti-HPV 31 | 100.0 [98.1 to 100.0]
  Anti-HPV 33: number analyzed (Participants) | 194
  Anti-HPV 33 | 100.0 [98.1 to 100.0]
  Anti-HPV 45: number analyzed (Participants) | 193
  Anti-HPV 45 | 100.0 [98.1 to 100.0]
  Anti-HPV 52: number analyzed (Participants) | 192
  Anti-HPV 52 | 100.0 [98.1 to 100.0]
  Anti-HPV 58: number analyzed (Participants) | 190
  Anti-HPV 58 | 100.0 [98.1 to 100.0]

2. Secondary Outcome: Percentage of Participants With a Solicited Injection-site Adverse Event
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant which did not necessarily have a causal relationship with study vaccine. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study vaccine or a protocol-specified procedure, whether or not considered related to the study vaccine or protocol-specified procedure. Any worsening of a preexisting condition that was temporally associated with the study vaccine or protocol-specified procedure was also an AE. The participant or the parent/guardian of the participant were to record the presence of any vaccination report card (VRC)-prompted injection-site AEs that occurred in the 5 days after any vaccination. The percentage of participants with an injection-site AE prompted on the VRC (erythema, pain, and swelling) was summarized.
Time Frame: Up to 5 days after any vaccination
Population: All participants that received at least 1 vaccination with 9vHPV vaccine and provided safety data at any time during the study.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 9vHPV Vaccine
Number analyzed (Participants) | 200
Percentage of Participants | 45.0 [38.0 to 52.2]

3. Secondary Outcome: Percentage of Participants With a Solicited Systemic Adverse Event
Description: An AE was defined as any untoward medical occurrence in a participant which did not necessarily have a causal relationship with study vaccine. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study vaccine or a protocol-specified procedure, whether or not considered related to the study vaccine or protocol-specified procedure. Any worsening of a preexisting condition that was temporally associated with the study vaccine or protocol-specified procedure was also an AE. The only solicited systemic AE was in response to results of daily oral temperature assessments. The participant or the parent/guardian of the participant will be asked to record the participant's oral temperature in the evening after each study vaccination and daily for 4 days after each study vaccination on VRC. The percentage of participants that had an AE due to an elevated oral temperature [(≥ 37.8 °C (100.0 °F)] was summarized.
Time Frame: Up to 5 days after any vaccination
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | 9vHPV Vaccine
Number analyzed (Participants) | 200
Percentage of Participants | 0.0

4. Secondary Outcome: Percentage of Participants With a Vaccine-related Serious Adverse Event
Description: A serious adverse event (SAE) is an AE that is life-threatening, requires or prolongs an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, or is another important medical event deemed such by medical or scientific judgment. The percentage of participants that experience at least one SAE that was reported as at least possibly related to the study vaccine was summarized.
Time Frame: Up to 4 weeks postdose 3 (Month 7)
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | 9vHPV Vaccine
Number analyzed (Participants) | 200
Percentage of Participants | 0.0

5. Secondary Outcome: Geometric Mean Titers of Serotype-specific Antibodies: Predose Day 1
Description: Anti-HPV Type 6, 11, 16, 18, 31, 33, 45, 52, and 58 antibodies are measured using a Competitive Luminex Immunoassay. Titers are reported in milli Merck units/mL (mMU/mL).
Time Frame: Day 1 (predose)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | 9vHPV Vaccine
Number analyzed (Participants) | 195
mMU/mL
  Anti-HPV 6: number analyzed (Participants) | 190
  Anti-HPV 6 | NA [NA to NA] — < Lower Limit of Quantification (LLOQ) of 20 mMU/mL
  Anti-HPV 11: number analyzed (Participants) | 190
  Anti-HPV 11 | NA [NA to NA] — < LLOQ of 16 mMU/mL
  Anti-HPV 16: number analyzed (Participants) | 187
  Anti-HPV 16 | NA [NA to NA] — < LLOQ of 20 mMU/mL
  Anti-HPV 18: number analyzed (Participants) | 190
  Anti-HPV 18 | 29.3 [27.7 to 31.1]
  Anti-HPV 31: number analyzed (Participants) | 188
  Anti-HPV 31 | NA [NA to NA] — < LLOQ of 10 mMU/mL
  Anti-HPV 33: number analyzed (Participants) | 194
  Anti-HPV 33 | NA [NA to 8.3] — < LLOQ of 8 mMU/mL
  Anti-HPV 45: number analyzed (Participants) | 193
  Anti-HPV 45 | NA [NA to NA] — < LLOQ of 8 mMU/mL
  Anti-HPV 52: number analyzed (Participants) | 192
  Anti-HPV 52 | NA [NA to NA] — < LLOQ of 8 mMU/mL
  Anti-HPV 58: number analyzed (Participants) | 190
  Anti-HPV 58 | NA [NA to NA] — < LLOQ of 8 mMU/mL

6. Secondary Outcome: Geometric Mean Titers of Antibodies to HPV 6, 11, 16, 18, 31, 33, 45, 52, and 58 at Month 7
Description: Anti-HPV Type 6, 11, 16, 18, 31, 33, 45, 52, and 58 antibodies are measured using a Competitive Luminex Immunoassay. Titers are reported in mMU/mL.
Time Frame: 4 weeks postdose 3 (Month 7)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Arm/Group | 9vHPV Vaccine
Number analyzed (Participants) | 195
mMU/mL
  Anti-HPV 6: number analyzed (Participants) | 190
  Anti-HPV 6 | 1008.2 [921.9 to 1102.6]
  Anti-HPV 11: number analyzed (Participants) | 190
  Anti-HPV 11 | 796.3 [722.2 to 878.0]
  Anti-HPV 16: number analyzed (Participants) | 187
  Anti-HPV 16 | 4605.4 [4163.7 to 5093.9]
  Anti-HPV 18: number analyzed (Participants) | 190
  Anti-HPV 18 | 1621.6 [1441.2 to 1824.5]
  Anti-HPV 31: number analyzed (Participants) | 188
  Anti-HPV 31 | 1137.9 [1017.2 to 1273.0]
  Anti-HPV 33: number analyzed (Participants) | 194
  Anti-HPV 33 | 507.8 [458.5 to 562.4]
  Anti-HPV 45: number analyzed (Participants) | 193
  Anti-HPV 45 | 579.2 [511.7 to 655.6]
  Anti-HPV 52: number analyzed (Participants) | 192
  Anti-HPV 52 | 500.8 [450.5 to 556.7]
  Anti-HPV 58: number analyzed (Participants) | 190
  Anti-HPV 58 | 701.8 [628.5 to 783.7]

ADVERSE EVENTS:
Time Frame: Up to 4 weeks postdose 3 (Month 7)
Description: Population for All-cause mortality included all enrolled participants. Population for Non-serious adverse events and serious adverse events included all participants that received at least 1 vaccination with 9vHPV vaccine and provided safety data at any time during the study.
Arm/Group | 9vHPV Vaccine
All-Cause Mortality (participants affected / at risk) | 0/201
Serious Adverse Events (participants affected / at risk) | 1/200
Other Adverse Events (participants affected / at risk) | 90/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 9vHPV Vaccine (N=200)
Subcutaneous abscess (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 9vHPV Vaccine (N=200)
Injection site pain (General disorders) | 89 (138)
Injection site swelling (General disorders) | 12 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the sponsor, the investigator agrees to submit all manuscripts or abstracts to the sponsor before submission. This allows the sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-19): https://cdn.clinicaltrials.gov/large-docs/42/NCT03546842/Prot_SAP_000.pdf